CLINICAL TRIAL: NCT01995305
Title: Exome Sequencing of Fanconi Anemia Children and the Their Parents
Brief Title: Use Massive Parallel Sequencing and Exome Capture Technology to Sequence the Exome of Fanconi Anemia Children and Their Patents
Status: Available | Type: Expanded Access
Sponsor: Xiaofan Zhu (Unknown)
Responsible Party: Sponsor-Investigator, Xiaofan Zhu, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Other Study IDs: pumc001; zhm001 (Other: pumc)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Fanconi Anemia; Autosomal or Sex Linked Recessive Genetic Disease; Bone Marrow Hematopoiesis Failure, Multiple Congenital Abnormalities, and Susceptibility to Neoplastic Diseases.; Hematopoiesis Maintainance.
Keywords: fanconi anemia; hematopoiesis maintainance
MeSH Terms: conditions — Fanconi Anemia; Abnormalities, Multiple | interventions — DNA Probes; Exome Sequencing

INTERVENTIONS:
Genetic: human whole exome — he exome is the part of the genome formed by exons, coding portions of genes in the genome that are used in the synthesis of proteins, therefore, it is most likely to contribute to the phenotype of an organism. The exome of the human genome, is estimated to comprise 1.5% of the total genome (The human exome is about 30 MB).
Genetic: whole genomic — This study propose to find the genes that are sensitive to DNA crosslink repair, and genes that have key roles in hematopoietic cell development and maturation.
  Other Names: whole exome

SUMMARY:
Fanconi anemia is a rare autosomal or sex linked recessive genetic disease. The disease is characterized by bone marrow hematopoiesis failure, multiple congenital abnormalities, and susceptibility to neoplastic diseases. The cells of FA patients are extremely sensitive to MMC and DEB. The symptoms and ages of FA patients are different, so by comparing the exome of FA patients and their parents, the mutations that were accumulated in FA patients could be found, and these genes might be sensitive to repairment and be important for hematopoiesis maintainance.

DETAILED DESCRIPTION:
Heterogeneity of FA. In the research of animal model, the phenotypes of FANCA, FANCC and FANCG knockout mice are similar. They grow up and develop normally, without any severe blood disease or tumor. However, they show chromosome instablity and highly sensitivity to MMC. And they have gonadal dysfunction and fertility defects. From this we conclude that the severe physical deformity of FA patients might be induced by other mutations. By comparing among the FA patients and between FA patiens and normal people, we look forward to find the mutated genes and verify their relationship with the physical deformity.

Even in 90% of FA patients the bone marrow failure will eventually occur, but the starting age ranges from 8-84. And Immuno-inhibition therapy has no effects on FA. Other DNA repair dysfunction diseases have higher rate of tumor, but not so high rate of bone marrow failure as FA does, which implies that the FA protein has the key role in hematopoietic stem cell maintainance. In FancC-/- mice, young mice is insensitive to DNA crosslinks with comet assay, but not adult mice, indicating that the accumulation of DNA damage during time leads to DNA repairment defects. by comparing the exome of FA patients and their parents, the mutations that were accumulated in FA patients could be found, and these genes might be sensitive to repairment and be important for hematopoiesis maintainance.

ELIGIBILITY:
Inclusion Criteria:

All the children that are diagnosed to be FA patients at the Blood Disease Hospital between 08/01/2010 - 07/31/2011, will be asked to participated in this study after acquiring the consent.

Exclusion Criteria:

Can not acquiring content

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tao Cheng, professor, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

REFERENCES:
- See also: informatin about this study — http://www.rockefeller.edu/fanconi/mutate